CLINICAL TRIAL: NCT07195630
Title: Both Acute Moderate-Intensity Continuous Exercise and High-Intensity Interval Exercise Increase Serum Oncostatin M Levels in Recreationally Active Males
Brief Title: Exercise-Induced Changes in Serum Oncostatin M Levels in Recreationally Active Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, İbrahim Türkel, LECTURER, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023/02-27
Record Dates: First submitted 2025-09-13; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: The Aim of This Study is to Evaluate the Effects of Acute Exercise on Serum Oncostatin M Levels in Healthy, Recreationally Active Males
Keywords: Acute Exercise; HIIT; Oncostatin M; MICE
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-intensity continuous exercise (MICE) (Experimental): 15 recreationally active males completed the ~21 min of exercise at 55% of VO2max, consisting of a 3-minute warm-up and 3-minute cool-down at 60 W.
  Interventions: Other: Moderate-Intensity Continuous Exercise
- High-intensity interval exercise (HIIE) (Experimental): 15 recreationally active males performed 10 x 1-minute intervals at 90% of VO2max, separated by 75 s of active recovery at 60 W, and a final 3-minute cool-down period at 60 W.
  Interventions: Other: High-Intensity Interval Exercise

INTERVENTIONS:
Other: Moderate-Intensity Continuous Exercise — 15 recreationally active males completed the ~21 min of exercise at 55% of VO2max, consisting of a 3-minute warm-up and 3-minute cool-down at 60 W.
  Arms: Moderate-intensity continuous exercise (MICE)
Other: High-Intensity Interval Exercise — 15 recreationally active males performed 10 x 1-minute intervals at 90% of VO2max, separated by 75 s of active recovery at 60 W, and a final 3-minute cool-down period at 60 W.
  Arms: High-intensity interval exercise (HIIE)

SUMMARY:
The aim of this study was to compare the effects of workload-matched acute moderate-intensity continuous exercise (MICE) and high-intensity interval exercise (HIIE) on serum OSM levels on a cycle ergometer in recreationally active, healthy men. Fifteen participants participated in both MICE and HIIE sessions. The HIIE session consisted of 10 x 1 min intervals at 90% of maximal oxygen uptake (VO2max) separated by a 75-second active recovery period at 60 W, whereas the MICE session consisted of a ~21 min exercise session at 55% of VO2max. Blood samples were collected before (Pre) and immediately after (Post) acute MICE and HIIE sessions. Serum OSM levels were measured by the ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Engaged in regular exercise/training in the last 6 months,
* 18-30 years of age,
* Body mass index (BMI) in the range of 18.5-24.9 kg/m².

Exclusion Criteria:

* Having a chronic disease that limits exercise,
* Smoking,
* Using any medication or supplement that may affect metabolism.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Change from Pre- to Post-Exercise Levels of Oncostatin M | From baseline assessment of blood samples at pre-exercise to the assessment of blood sample analysis at the end of the post-exercise.
  Serum samples were collected at pre- and post-exercise time points, and serum oncostatin M levels were measured using a commercial ELISA kit

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No